CLINICAL TRIAL: NCT06219460
Title: A Comparison of Two Types of Face Masks: Cuffed and Uncuffed for Ventilation of Obese Patients
Brief Title: Comparison of Two Types of Face Mask Ventilation in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Tomasz Gaszynski, prof. dr hab., Medical University of Lodz
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RNN/96/13/KB
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Morbid
Keywords: morbid obesity; face mask ventilation
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cuffed face amsk (Experimental): Ventilation using cuffed face mask
  Interventions: Other: Ventilation using two types of face masks
- Uncuffed face mask (Experimental): Ventilation using uncuffed face mask
  Interventions: Other: Ventilation using two types of face masks

INTERVENTIONS:
Other: Ventilation using two types of face masks — ventilation using two types of face mask

SUMMARY:
Two types of face masks : cuffed and uncuffed were evaluated for artificial ventilation in obese patients. After induction to anesthesia patients were ventilated with both types of masks using anesthesia machine with the same settings: Tital Volume of 500 ml, respiratory rate of 12/min. The inspired and expired volume was measured using anesthesia machine volumeter, The difference between inspired and expired volume was counted. The comparison between two types of masks was performed taking into consideration several parameters: type of obesity, gender, age.

DETAILED DESCRIPTION:
The aim of the study was to determine which of the tested: cuffed or uncuffed face masks allows better replacement ventilation in obese patients.

The study was conducted on patients with the BMI over 39 kg/m2 Patients qualified for bariatric surgery were selected for this study according to the order of reporting to the surgery department. The study adopted a simplified assumption that the gynoid type of obesity most often concerns women, and the android type, i.e. abdominal obesity, most often affects men. Two face masks were used to compare the effectiveness of replacement ventilation: the cuffed and uncuffed . It was randomly chosen (by tossing a coin) which face mask would be used first. The induction of anesthesia was low-opioid, the patients were placed in the supine position with the head and trunk elevated by 25 degrees on a positioning pad. 100% oxygen concentration was used for active pre-oxygenation, the test mask was applied with one hand using the EC clamp technique. The masks were changed after four consecutive measurements for each type of mask. In order to objectify the measurement with the same tidal volume, a respirator was used with the same settings: Tidal Volume of 500 ml and respiratory rate of 12/min. Sealing was measured by comparing the inspired volume with expired volume, that is the amount of leakage generated by individual masks was assessed. The obtained data were analyzed with the Kolmogorow-Smirnov test and supplemented with the values of the Wilcoxona test.

ELIGIBILITY:
Inclusion Criteria:

* obesity
* scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* predicted difficult intubation
* predicted difficult face-mask ventilation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Sealing of face masks measured by difference of inspired tidal volume and expired volume | immediatethrough study completion
  Sealing of cuffed or uncuffed masks during face mask ventilation in obese patients measred by anesthesia machine

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Gaszynski, Prof, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No